CLINICAL TRIAL: NCT01326247
Title: EFFECTIVENESS OF THERAPY WITH A THERMAL WATER NASAL AEROSOL IN CHILDREN WITH SEASONAL ALLERGIC RHINITIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Collaborators: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Michele Miraglia del Giudice, MD, Dipartimento di Pediatria "F.Fede" - Seconda Università di Napoli
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: studioterme
Record Dates: First submitted 2011-03-28; First posted 2011-03-30 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2009-12

CONDITIONS: Allergic Rhinitis (Disorder)
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 0.9% NaCl solution (No Intervention)
  Interventions: Other: thermal waters nasal irrigation

INTERVENTIONS:
Other: thermal waters nasal irrigation — The first group (group 1) has practiced crenotherapy with "hyper-mineral chloride sodium water" aerosol by nasal adapter for 15 days per month, for three consecutive months, at thermal spa services of Lacco Ameno, while the control group (group 2) was treated, in the same period, daily, by a micronized nasal douche with 0.9% NaCl (isotonic) solution.

SUMMARY:
The purpose of this study was to evaluate the effects of Ischia thermal waters nasal irrigation on allergic rhinitis and airway inflammation during the period of natural exposure to parietaria pollen in children with allergic rhinitis and intermittent asthma.

DETAILED DESCRIPTION:
The study was conducted on the island of Ischia - Naples from April to June 2009, during the natural exposure period to parietaria pollen. The treatment started just before the pollen season, when all the children were asymptomatic, not treated with any drug and not affected by respiratory tract and systemic diseases. All the children were randomly divided into two homogeneous groups by sex and age. The first group has practiced crenotherapy with "hyper-mineral chloride sodium water" aerosol by nasal adapter for 15 days per month, for three consecutive months, at thermal spa services of Lacco Ameno, while the control group was treated, in the same period, daily, by a micronized nasal douche with 0.9% NaCl (isotonic) solution. Before the treatment (T0), at the end of the treatment (T1) and again 2 weeks after the end of the treatment (T2), all the children have performed spirometry (Pony FX Cosmed), and exhaled nitric oxide (FeNO) (NIOX MINO analyzer COSMED), to assess their airway inflammation. At the time of recruitment, the parents of the children were instructed to fill a specific diary-card (TSS) at home, to assess rhinitis symptoms and possible drug use during all 3 months of treatment. The parameters considered in the TSS were: nasal obstruction, sneezing, nasal discharge and itching. These symptoms were scored: 0 = symptom absent, 1 = mild (symptoms present but not annoying), 2 = moderate (frequent and offensive symptoms but do not interfere with sleep or normal activities) 3 = severe (symptoms that interfere with sleep or normal activities).

Every two weeks, at the end of each cycle of therapy the children underwent a general clinical control with nasal endoscopy, spirometry and monitoring the completion of diary cards and the possible use of drugs.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of moderate to severe allergic rhinitis.
* Children aged 6-14 year sensitized to parietaria.
* History of spring time symptoms.
* History of mild intermittent asthma.

Exclusion Criteria:

* Use of LABA, antihistamines, intranasal, bronchial or systemic corticosteroids, cromolyn sodium and leukotriene modifiers in the last 6 weeks.
* The presence of respiratory tract infection, persistent asthma, respiratory tract abnormalities or diseases.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The Primary Outcome was to measure the differences in nasal symptoms score (TSS) about groups after three months of therapy. Data were compared by the Mann-Whitney test.
  At the time of recruitment, the parents of the children were instructed to fill a specific diary-card (TSS) at home, to assess rhinitis symptoms and possible drug use during all 3 months of treatment. The parameters considered in the TSS were: nasal obstruction, sneezing, nasal discharge and itching. These symptoms were scored: 0 = symptom absent, 1 = mild (symptoms present but not annoying), 2 = moderate (frequent and offensive symptoms but do not interfere with sleep or normal activities) 3 = severe (symptoms that interfere with sleep or normal activities).

SECONDARY OUTCOMES:
exhaled nitric oxide (FeNO) by NIOX MINO analyzer COSMED, to assess airway inflammation.
  It's well known that allergic rhinitis is often associated with asthma. Allergic rhinitis and asthma are expressions of respiratory mucosal eosinophilic inflammation. Before the treatment (T0), at the end of the treatment (T1) and again 2 weeks after the end of the treatment (T2), all the children have performed spirometry and exhaled nitric oxide (FeNO) (NIOX MINO analyzer COSMED), to assess their airway inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Miraglia del Giudice, MD, Principal Investigator — Dipartimento di Pediatria "F.Fede" - Seconda Università di Napoli
Locations (1):
- UOC Pediatria e Neonatologia, ASL Na-2, PO "Anna Rizzoli", Ischia, Campania, Italy

REFERENCES:
- [Derived] Miraglia Del Giudice M, Decimo F, Maiello N, Leonardi S, Parisi G, Golluccio M, Capasso M, Balestrieri U, Rocco A, Perrone L, Ciprandi G. Effectiveness of Ischia thermal water nasal aerosol in children with seasonal allergic rhinitis: a randomized and controlled study. Int J Immunopathol Pharmacol. 2011 Oct-Dec;24(4):1103-9. doi: 10.1177/039463201102400431. PMID 22230419